CLINICAL TRIAL: NCT07154459
Title: A Study to Assess the Impact of Breastfeeding Education on Prenatal and Paternal Attachment in Primiparous Parents
Brief Title: Breastfeeding Education and Prenatal & Paternal Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gizem ÇITAK (Other)
Collaborators: Tokat Gaziosmanpasa University (Other)
Responsible Party: Sponsor-Investigator, Gizem ÇITAK, Asist. Prof. Dr., Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: K21.28
Record Dates: First submitted 2025-07-22; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Prenatal Attachment; Paternal Behavior; Pregnancy; Breastfeeding
Keywords: Prenatal attachment; Paternal Behavior; Pregnancy; Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): Breastfeeding education group
  Interventions: Other: Breastfeeding Education
- Control (No Intervention): Non-education group

INTERVENTIONS:
Other: Breastfeeding Education — Breastfeeding Education
  Arms: Education

SUMMARY:
This study is designed to evaluate the effect of breastfeeding education on prenatal attachment and paternal attachment among first-time parents. A total of 101 first-time parents (52 in the intervention group and 49 in the control group) will be recruited. Pregnant women will complete the Prenatal Attachment Inventory before and after the intervention, and expectant fathers will complete the Paternal Prenatal Attachment Inventory before and after the intervention. Participants will be selected using non-probability and snowball sampling methods, and the breastfeeding education will be delivered online via Google Meet. The study aims to assess whether structured breastfeeding education can influence prenatal and paternal attachment in first-time parents.

DETAILED DESCRIPTION:
Background: Breastfeeding education is recognized as an important factor supporting mother-infant bonding. However, there is limited research on the impact of such education on prenatal bonding for both mothers and fathers, especially among first-time parents (primiparous). Understanding how breastfeeding education influences prenatal attachment in this group is crucial for enhancing parental bonding and early family health.

Aim: This study aims to evaluate the effect of breastfeeding education on prenatal bonding in primiparous parents, focusing on both maternal and paternal attachment.

Method: A total of 101 primiparous parents participated in the study, with 52 in the experimental group and 49 in the control group. Pregnant women completed the Prenatal Attachment Scale before and after receiving breastfeeding education, while expectant fathers completed the Paternal Antenatal Attachment Scale pre- and post-education. Participants were recruited using non-probability and snowball sampling methods, and the education sessions were delivered online via Google Meet.

ELIGIBILITY:
Inclusion Criteria:• Primiparous pregnant women

* Age 20 years or older
* In the second or third trimester of pregnancy
* Having internet access

Exclusion Criteria Not being a primiparous pregnant woman

* Under 20 years of age
* Refusal or withdrawal from the education or data collection process
* Withdrawal from the study before completing the education
* Incomplete pre-test or post-test data
* Non-compliance with the study protocol

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Prenatal Attachment | 4 Week
  Measuring prenatal attachment through breastfeeding education using the Prenatal Attachment Scale; scores range from 1 to 5, with higher scores indicating stronger attachment.

SECONDARY OUTCOMES:
Paternal Attachment | 4 week
  Measuring paternal attachment through breastfeeding education using the Paternal Antenatal Attachment Scale; scores range from 1 to 5, with higher scores indicating stronger attachment.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem ÇITAK, Asst Prof, Principal Investigator — Tokat Gaziosmanpaşa University
Locations (1):
- Tokat Gaziosmanpaşa University Rectorate General Secretariat Taşlıçiftlik Campus, 60250 Tokat/Central, Tokat Province, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to participant confidentiality and ethical regulations.